CLINICAL TRIAL: NCT03009916
Title: Bileacid Malabsorption and GLP-1 Secretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-15004394
Record Dates: First submitted 2016-12-21; First posted 2017-01-04 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Bileacid Malabsorption
MeSH Terms: interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Healthy controls (Other): Healthy controls found according to the protocol
  Interventions: Drug: "cholestagel®" (Colesevelam); Drug: Placebos
- Patients with BAM (Other): Patients with bile acid malabsorption found according to the protocol
  Interventions: Drug: "cholestagel®" (Colesevelam); Drug: Placebos

INTERVENTIONS:
Drug: "cholestagel®" (Colesevelam) — 3750mg
Drug: Placebos — 3750mg

SUMMARY:
The aim of this study is to examine the influence of BAM on postprandial GLP--1 secretion and glucose homeostasis, both with and without bile acid sequestration.

ELIGIBILITY:
Inclusion Criteria:

* Northern European origin
* Normal haemoglobin
* Age above 18 years and below 70 years
* Informed and written consent
* BMI > 23 kg/m2 and < 35 kg/m2
* Normal fasting plasma glucose (FPG) < 6.5 mM) and glycated haemoglobin (HbA1c) < 48 mmol/mol

Exclusion Criteria:

* Liver disease (alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder
* Gastrointestinal disease (except BAM), previous intestinal resection, cholecystectomy or any major intra-abdominal surgery
* First-degree relatives with diabetes
* Nephropathy (serum creatinine >150 µM and/or albuminuria
* Treatment with medicine that cannot be paused for 12 hours
* Hypothyroidism or hyperthyroidism
* Treatment with oral anticoagulants
* Active or recent malignant disease
* Any treatment or condition requiring acute or sub-acute medical or surgical intervention
* Lack of effective birth control in premenopausal women
* Any condition considered incompatible with participation by the investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
GLP-1 | 240 min

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Karhus ML, Sonne DP, Thomasen M, Ellegaard AM, Holst JJ, Rehfeld JF, Chavez-Talavera O, Tailleux A, Staels B, Nielsen DS, Krych L, Dragsted LO, Vilsboll T, Bronden A, Knop FK. Enterohepatic, Gluco-metabolic, and Gut Microbial Characterization of Individuals With Bile Acid Malabsorption. Gastro Hep Adv. 2022 Mar 30;1(3):299-312. doi: 10.1016/j.gastha.2021.12.007. eCollection 2022. PMID 39131668